CLINICAL TRIAL: NCT01863771
Title: A Phase 3 Multicenter, Placebo-controlled, Double-blind, Randomized-withdrawal Study to Evaluate the Safety and Efficacy of Golimumab Maintenance Therapy, Administered Subcutaneously, in Japanese Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Safety and Effectiveness Study of Golimumab in Japanese Patients With Moderately to Severely Active Ulcerative Colitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100937; CNTO148UCO3001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Colitis, Ulcerative
Keywords: Ulcerative Colitis; Japanese; Subcutaneous; Golimumab
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Golimumab (Experimental)
  Interventions: Drug: Golimumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Golimumab — Participants will receive 200 mg golimumab at Week 0 and 100 mg golimumab at Week 2 as a subcutaneous (SC) (under the skin) injection in the induction phase. Participants who have a clinical response in the induction phase and are randomly allocated to golimumab in the maintenance phase will receive 100 mg SC every 4 weeks through Week 52. Participants who do not have a clinical response in the induction phase will receive 100 mg of golimumab SC at Week 4 and will continue with 100 mg of golimumab SC every 4 weeks through Week 52 only if a response is obtained by Week 8.
  Arms: Golimumab
Other: Placebo — Participants who have a clinical response to golimumab in the induction phase and are randomly allocated to placebo in the maintenance phase will receive SC placebo every 4 weeks through Week 52. However, participants receiving placebo and who will lose clinical response any time during the study will be eligible to receive 100 mg golimumab SC every 4 weeks through Week 52.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and effectiveness of golimumab in Japanese participants with moderately to severely active ulcerative colitis.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (study in which an inactive substance is given to one group of participants, while the study medication is given to another group), multicenter (study conducted at multiple sites), 2-arm (two groups), parallel-group (each group of participants will be treated at the same time), randomized-withdrawal (participants receiving study medication for a specified time will be later randomized to receive either study medication or placebo.) study, including an open-label (all people know the identity of the intervention) induction phase. Approximately 200 participants will participate in this study. This study will consist of an induction phase, a maintenance phase, and a follow-up phase. During the induction phase (lasting 6 weeks) participants will receive 200 mg subcutaneous (SC) (under the skin) golimumab at Week 0 and 100 mg SC golimumab at Week 2. During the maintenance phase (up to Week 52) all participants who show a clinical response (measure of therapeutic effect of study medication) to golimumab during the induction phase will be randomly allocated in a 1:1 ratio to receive either SC administration of placebo (Group 1) or 100 mg golimumab (Group 2) every 4 weeks from Week 0 to Week 52. Participants who do not show clinical response to golimumab will also receive 100 mg SC administration of golimumab until Week 4 and if, by Week 8 of the maintenance phase, these participant's disease activity does not appear to be improving, participants will be discontinued from further study medication administration and will be followed up for safety evaluations 16 weeks after the last administration of study medication. However, if disease activity of these participants improves at Week 8, they will continue to receive golimumab (100 mg every 4 weeks) through Week 52 of the maintenance phase. The follow-up phase will be of 16 weeks duration. During this study, any participant who have a clinical response during the induction phase but lose clinical response at any time will be eligible for dose adjustment only once as follows: 1) participants receiving placebo (Group 1) will receive golimumab 100 mg; 2) participants receiving golimumab 100 mg (Group 2) will continue to receive golimumab 100 mg. Safety evaluations will include assessment of adverse events, laboratory measurements, antinuclear antibodies/anti-double-stranded deoxyribonucleic acid antibodies, and vital signs. The maximum study duration for a participant will be 68 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ulcerative colitis diagnosed prior to screening
* Participants should have current treatment for ulcerative colitis with at least one of the following therapies: oral 5-aminosalicylates (5-ASAs), oral corticosteroids, 6-mercaptopurine (6-MP), or azathioprine (AZA)
* Participants must have a history of failure to respond to, or tolerate, at least 1 of the following therapies: oral 5-ASAs, oral corticosteroids, 6-MP, or AZA
* Participants must be ambulatory and have moderately to severely active ulcerative colitis confirmed during the screening sigmoidoscopy by a greater than or equal to 2 using the endoscopy subscore of the Mayo score
* Participants must have moderately to severely active ulcerative colitis, defined as a baseline Mayo score of 6 to 12, inclusive

Exclusion Criteria:

* Participants with ulcerative colitis limited to the rectum only or to less than 20 cm of the colon
* Participants with stoma
* Participants with fistula or history of fistula
* Participants who require, or required within the 2 months prior to screening, surgery for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage, or other conditions possibly confounding the evaluation of benefit from study agent treatment
* Participants with symptomatic colonic or small bowel obstruction, confirmed by objective radiographic or endoscopic evidence of a stricture with resulting obstruction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2016-01-29 (Actual); Study Completion 2016-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (38):
- Japan (38):
  - Abiko
  - Chiba
  - Chikushinoshi
  - Fujiidera
  - Fukuoka
  - Fushimi
  - Hamamatsu
  - Hirosaki
  - Hiroshima
  - Ikeda
  - Izumiōtsu
  - Izumo
  - Kagoshima
  - Kahoku
  - Kanazawa
  - Kochi
  - Kurume
  - Maebashi
  - Miyazaki
  - Nagasaki
  - Nagoya
  - Nishinomiya
  - Osaka
  - Ōita
  - Saga
  - Sakura
  - Sapporo
  - Sendai
  - Suita
  - Sunto
  - Tokushima
  - Tokyo
  - Toyota
  - Tsu
  - Tsukuba
  - Wakayama
  - Yokkaichi
  - Yokohama

REFERENCES:
- [Derived] Hibi T, Imai Y, Senoo A, Ohta K, Ukyo Y. Efficacy and safety of golimumab 52-week maintenance therapy in Japanese patients with moderate to severely active ulcerative colitis: a phase 3, double-blind, randomized, placebo-controlled study-(PURSUIT-J study). J Gastroenterol. 2017 Oct;52(10):1101-1111. doi: 10.1007/s00535-017-1326-1. Epub 2017 Mar 21. PMID 28324167

RESULTS

PARTICIPANT FLOW:
Groups:
- Group1: Golimumab [Induction]: Participants received golimumab 200 milligram (mg) once at Week 0 and golimumab 100 mg once at Week 2 subcutaneously (SC).
- Group 2: Golimumab 100 mg [Maintenance]: Participants who responded to golimumab induction treatment received golimumab 100 mg SC every 4 weeks (q4w) through Week 52.
- Group 3: Placebo [Maintenance]: Participants who responded to golimumab induction treatment received placebo SC every 4 weeks (q4w) through Week 52.
- Group 4: Golimumab 100 mg [Maintenance]: Participants who not responded to golimumab induction dosing received golimumab 100 mg SC once at Week 0 and once at Week 4, and based on clinical response every 4 weeks through Week 52.
Period: Induction Phase
Arm/Group | Group1: Golimumab [Induction] | Group 2: Golimumab 100 mg [Maintenance] | Group 3: Placebo [Maintenance] | Group 4: Golimumab 100 mg [Maintenance]
Started | 144 | 0 | 0 | 0
Completed | 123 (Same participants who completed the induction phase participated in the maintenance phase.) | 0 | 0 | 0
Not Completed | 21 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Group1: Golimumab [Induction] | Group 2: Golimumab 100 mg [Maintenance] | Group 3: Placebo [Maintenance] | Group 4: Golimumab 100 mg [Maintenance]
Started | 0 | 32 | 31 | 60
Completed | 0 | 27 | 19 | 17
Not Completed | 0 | 5 | 12 | 43
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 3 | 7 | 38
Not completed — Physician Decision | 0 | 0 | 2 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Efficacy full analysis set for induction phase (FAS-I) included all participants who were treated in the induction phase.
Groups:
- All Participants: Participants who received golimumab 200 milligram (mg) once at Week 0 and golimumab 100 mg once at Week 2 subcutaneously (SC) in the induction phase.
Arm/Group | All Participants
Number analyzed (Participants) | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 98
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Clinical Response Through Maintenance-Week 54 Measured Using the Mayo Score
Description: Clinical response was defined as a decrease from Induction-Week 0 in the Mayo score by greater than or equal to (>=) 30 percent and >=3 points, with a decrease in the rectal bleeding subscore of >= 1 or a rectal bleeding subscore of 0 or 1. The Mayo score is the primary tool for assessing ulcerative colitis activity. The Mayo score consists of 4 subscores (stool frequency, rectal bleeding, findings of endoscopy, and physician's global assessment) which range from 0 to 3. The Mayo score is calculated as the sum of these 4 subscores and can range between 0 and 12. A score of 3 to 5 points indicates mildly active disease; a score of 6 to 10 indicates moderately active disease; and a score of 11 to 12 indicates severe disease.
Time Frame: Up to Week 54
Population: Efficacy full analysis set for maintenance phase included all participants who responded to golimumab induction treatment and subsequently randomized at Week 0 in maintenance phase. Data for this outcome was not planned to be analyzed for participants who had not responded to golimumab induction dosing, as pre-specified in protocol.
Measure: Number; unit: participants
Groups:
- Placebo: Participants who responded to golimumab induction treatment received placebo subcutaneously (SC) every 4 weeks (q4w) through Week 52 in the maintenance phase.
- Golimumab: Participants received golimumab 200 mg (once at Week 0) and golimumab 100 mg (once at Week 2) SC in induction phase. Participants who responded to golimumab induction treatment received golimumab 100 mg SC, q4w through Week 52 and participants who not responded to golimumab induction treatment received golimumab 100 mg SC at Weeks 0 and 4, and based on clinical response every 4 weeks through Week 52 in maintenance phase.
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 31 | 32
participants | 6 [5.4 to 33.3] | 18 [39.1 to 73.4]

2. Secondary Outcome: Number of Participants Who Achieved Clinical Remission at Both Maintenance-Week 30 and Week 54
Description: Clinical remission (as measured by the Mayo score) was defined as a Mayo score of less than or equal to (<=) 2 points, with no individual sub-score greater than (>) 1.
Time Frame: Weeks 30 and 54
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 31 | 32
participants | 2 | 16

3. Secondary Outcome: Number of Participants With Mucosal Healing at Both Maintenance-Week 30 and Week 54
Description: Mucosal healing is defined as an endoscopy subscore of 0 or 1, where 0 indicates normal or inactive disease and 1 indicates mild disease (erythema, decreased vascular pattern, mild friability). Endoscopy subscore is one of the 4 subscores of the Mayo score.
Time Frame: Weeks 30 and 54
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Golimumab
Number analyzed (Participants) | 31 | 32
participants | 5 | 19

ADVERSE EVENTS:
Description: Safety data were analyzed separately for all treated participants in the induction phase and randomized and non-randomized participants in the maintenance phase. Participants were analyzed according to the actual treatment they received.
Groups:
- Group 4: Golimumab 100 mg [Maintenance]: Participants who not responded to golimumab induction dosing received golimumab 100 mg SC once at Week 0 and once at Week 4, and based on clinical response every 4 week through Week 52.
Arm/Group | Group1: Golimumab [Induction] | Group 2: Golimumab 100 mg [Maintenance] | Group 3: Placebo [Maintenance] | Group 4: Golimumab 100 mg [Maintenance]
Serious Adverse Events (participants affected / at risk) | 5/144 | 1/32 | 4/31 | 6/60
Other Adverse Events (participants affected / at risk) | 36/144 | 26/32 | 15/31 | 31/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group1: Golimumab [Induction] (N=144) | Group 2: Golimumab 100 mg [Maintenance] (N=32) | Group 3: Placebo [Maintenance] (N=31) | Group 4: Golimumab 100 mg [Maintenance] (N=60)
Colitis Ulcerative (Gastrointestinal disorders) | 4 | 0 | 1 | 5
Cytomegalovirus Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Takayasu's Arteritis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group1: Golimumab [Induction] (N=144) | Group 2: Golimumab 100 mg [Maintenance] (N=32) | Group 3: Placebo [Maintenance] (N=31) | Group 4: Golimumab 100 mg [Maintenance] (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 7 | 0 | 2 | 4
Injection Site Erythema (General disorders) | 5 | 5 | 0 | 1
Injection Site Pain (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 4 | 1 | 3
Nasopharyngitis (Infections and infestations) | 17 | 17 | 7 | 14
Oral Herpes (Infections and infestations) | 0 | 1 | 3 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 2 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Headache (Nervous system disorders) | 3 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.